CLINICAL TRIAL: NCT04041570
Title: A Phase I Open-Label, Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of Two Doses of an Ebola Sudan Chimpanzee Adenovirus Vector Vaccine, VRC-EBOADC086-00-VP (cAd3-EBO S), in Healthy Adults
Brief Title: Ebola Sudan Chimpanzee Adenovirus Vector Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: US Military HIV Research Program (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RV 508; WRAIR 2439 (Other: WRAIR)
Record Dates: First submitted 2019-07-25; First posted 2019-08-01 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Ebola Virus
Keywords: Ebola virus; Ebola vaccine; cAd3-EBO S

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Dose Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: cAd3-EBO S vaccine (1x10^10 PU) (Experimental): cAd3-EBO S vaccine (1x10^10 PU) administered intramuscularly (IM) with needle and syringe in a volume of 1 mL
  Interventions: Biological: cAd3-EBO S vaccine
- Group 2: cAd3-EBO S vaccine (1x10^11 PU) (Experimental): cAd3-EBO S vaccine (1x10^11 PU) administered IM with needle and syringe in a volume of 1 mL
  Interventions: Biological: cAd3-EBO S vaccine

INTERVENTIONS:
Biological: cAd3-EBO S vaccine — The recombinant chimpanzee adenovirus Type 3-vectored Ebola vaccine, VRC-EBOADC086-00-VP (cAd3-EBO S), is composed of a cAd3 vector that encodes Ebola Sudan wild type glycoprotein (WT GP).
  Other Names: VRC-EBOADC086-00-VP

SUMMARY:
RV 508 was a Phase I, open-label, dose-escalation study to examine the safety, tolerability and immunogenicity of an investigational Ebola vaccine in healthy adults. VRC-EBOADC086-00-VP, a chimpanzee adenovirus serotype 3 vector-based Ebola vaccine, encodes wild type (WT) glycoprotein (GP) from the Sudan strain of Ebolavirus and is administered intramuscularly (IM).

DETAILED DESCRIPTION:
A total of 40 participants were evenly split, with 20 in each of the two dosage groups to receive the investigational cAd3-EBO S vaccine at a dose of either 1x10^10 particle units (PU) (Group 1) or 1x10^11 PU (Group 2). The dose escalation plan included daily review of any new safety data by a study clinician, regular review of safety data by the protocol team and a staged enrollment plan with required interim safety reviews. The study began with enrollment of 3 participants into Group 1 (1x10^10 PU) at a rate of 1 participant per day. After at least 7 days of follow-up for the first 3 vaccinated participants, an interim safety review occurred before enrollment of additional participants into the group. No safety issues were identified; therefore, an additional 17 participants were enrolled to complete Group 1. When there was a minimum of seven days of follow-up safety data from the last enrolled participant in Group 1, an interim safety review occurred. No safety issues were identified, and enrollment of participants into the next dose level (Group 2) began with the enrollment of 3 participants at a rate of 1 participant per day. After at least 7 days of follow-up for the first 3 vaccinated participants in Group 2 (1x10^11 PU), an interim safety review occurred before the enrollment of additional participants into Group 2. No safety issues were identified, and an additional 17 participants were enrolled to complete Group 2. Participants were followed for approximately 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 50 years old.
2. Available for clinical follow-up through Week 48 after enrollment.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Able and willing to provide fingerprints and have their photographs taken including injection site photographs.
5. Must allow home visits
6. Must complete an Assessment of Understanding (AoU) prior to enrollment by answering 9 out of 10 questions at least once in 3 attempts.
7. Able to read (English or Luganda) and willing to complete the informed consent process.
8. In good general health without clinically significant medical history.
9. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) ≤ 40 within the 56 days prior to enrollment.
10. Laboratory Criteria within 56 days prior to enrollment:

    1. Hemoglobin ≥ 11.0 g/dL for women; ≥12.5 g/dL for men.
    2. White blood cells (WBC) = 2,500-12,000 cells/mm^3.
    3. Total lymphocyte count ≥ 800 cells/mm^3.
    4. Platelets = 125,000 - 400,000/mm^3.
    5. Alanine aminotransferase (ALT) ≤ 1.25 x upper limit of normal.
    6. Serum creatinine ≤ 1 x upper limit of normal.
    7. HIV-uninfected as evidenced by a negative FDA-approved HIV diagnostic test.

    Female-Specific Criteria:
11. Negative β-HCG (human chorionic gonadotropin) pregnancy test; serum β-HCG at screening and urine β-HCG at enrollment if woman is of reproductive potential.
12. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 24 weeks after study vaccination if assessed to be of reproductive potential.

Exclusion Criteria:

Volunteer has received any of the following substances:

1. Investigational Ebola or Marburg vaccine in a prior clinical trial or prior receipt of a cAd3 adenoviral vectored investigational vaccine.
2. Chronic use of immunomodulators and systemic glucocorticoids in daily doses of glucocorticoid equivalence > 20 mg of prednisolone, for periods exceeding 10 days. Non-steroidal anti-inflammatory drugs [NSAIDS] are permitted. Participants that have used less than the stated glucocorticoid dose may still be excluded at the Investigator's discretion.
3. Blood products within 112 days (16 weeks) prior to enrollment.
4. Investigational research agents within 28 days (4 weeks) prior to enrollment.
5. Live attenuated vaccines within 28 days (4 weeks) prior to enrollment.
6. Subunit or killed vaccines within 14 days (2 weeks) prior to enrollment.
7. Current anti-tuberculosis prophylaxis or therapy.

   Female-specific criteria:
8. Woman who is pregnant, breast-feeding or planning to become pregnant during the first 24 weeks after study vaccine administration.

   Volunteer has a history of any of the following clinically significant conditions:
9. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
10. Allergic reaction to excipients in the study vaccine including gentamycin, neomycin or streptomycin.
11. Clinically significant autoimmune disease or immunodeficiency.
12. Asthma that is not well controlled.
13. Positive result on a rapid plasma reagin (RPR) test.
14. Diabetes mellitus (type I or II).
15. Thyroid disease that is not well controlled.
16. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
17. Idiopathic urticaria within the last 1 year.
18. Hypertension that is not well controlled.
19. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
20. A malignancy that is active, currently being treated, or not surgically cured.
21. Seizure in the past 3 years or treatment for seizure disorder in the past 3 years.
22. Asplenia or functional asplenia.
23. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within five years prior to enrollment, history of a suicide plan or attempt.
24. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University-Walter Reed Project, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarwar UN, Costner P, Enama ME, Berkowitz N, Hu Z, Hendel CS, Sitar S, Plummer S, Mulangu S, Bailer RT, Koup RA, Mascola JR, Nabel GJ, Sullivan NJ, Graham BS, Ledgerwood JE; VRC 206 Study Team. Safety and immunogenicity of DNA vaccines encoding Ebolavirus and Marburgvirus wild-type glycoproteins in a phase I clinical trial. J Infect Dis. 2015 Feb 15;211(4):549-57. doi: 10.1093/infdis/jiu511. Epub 2014 Sep 14. PMID 25225676
- [Background] Kibuuka H, Berkowitz NM, Millard M, Enama ME, Tindikahwa A, Sekiziyivu AB, Costner P, Sitar S, Glover D, Hu Z, Joshi G, Stanley D, Kunchai M, Eller LA, Bailer RT, Koup RA, Nabel GJ, Mascola JR, Sullivan NJ, Graham BS, Roederer M, Michael NL, Robb ML, Ledgerwood JE; RV 247 Study Team. Safety and immunogenicity of Ebola virus and Marburg virus glycoprotein DNA vaccines assessed separately and concomitantly in healthy Ugandan adults: a phase 1b, randomised, double-blind, placebo-controlled clinical trial. Lancet. 2015 Apr 18;385(9977):1545-54. doi: 10.1016/S0140-6736(14)62385-0. Epub 2014 Dec 23. PMID 25540891
- [Background] Ledgerwood JE, DeZure AD, Stanley DA, Coates EE, Novik L, Enama ME, Berkowitz NM, Hu Z, Joshi G, Ploquin A, Sitar S, Gordon IJ, Plummer SA, Holman LA, Hendel CS, Yamshchikov G, Roman F, Nicosia A, Colloca S, Cortese R, Bailer RT, Schwartz RM, Roederer M, Mascola JR, Koup RA, Sullivan NJ, Graham BS; VRC 207 Study Team. Chimpanzee Adenovirus Vector Ebola Vaccine. N Engl J Med. 2017 Mar 9;376(10):928-938. doi: 10.1056/NEJMoa1410863. Epub 2014 Nov 26. PMID 25426834
- [Background] Paris R, Kuschner RA, Binn L, Thomas SJ, Colloca S, Nicosia A, Cortese R, Bailer RT, Sullivan N, Koup RA. Adenovirus type 4 and 7 vaccination or adenovirus type 4 respiratory infection elicits minimal cross-reactive antibody responses to nonhuman adenovirus vaccine vectors. Clin Vaccine Immunol. 2014 May;21(5):783-6. doi: 10.1128/CVI.00011-14. Epub 2014 Mar 12. PMID 24623627
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1. [July 2017]. Available from: https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- [Background] Amai M, Nojima M, Yuki Y, Kiyono H, Nagamura F. A review of criteria strictness in "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". Vaccine. 2023 Aug 31;41(38):5622-5629. doi: 10.1016/j.vaccine.2023.07.072. Epub 2023 Aug 1. PMID 37532612
- [Derived] Mwesigwa B, Houser KV, Hofstetter AR, Ortega-Villa AM, Naluyima P, Kiweewa F, Nakabuye I, Yamshchikov GV, Andrews C, O'Callahan M, Strom L, Schech S, Anne Eller L, Sondergaard EL, Scott PT, Amare MF, Modjarrad K, Wamala A, Tindikahwa A, Musingye E, Nanyondo J, Gaudinski MR, Gordon IJ, Holman LA, Saunders JG, Costner PJM, Mendoza FH, Happe M, Morgan P, Plummer SH, Hickman SP, Vazquez S, Murray T, Cordon J, Dulan CNM, Hunegnaw R, Basappa M, Padilla M, Gajjala SR, Swanson PA 2nd, Lin BC, Coates EE, Gall JG, McDermott AB, Koup RA, Mascola JR, Ploquin A, Sullivan NJ, Kibuuka H, Ake JA, Ledgerwood JE; RV 508 Study Team. Safety, tolerability, and immunogenicity of the Ebola Sudan chimpanzee adenovirus vector vaccine (cAd3-EBO S) in healthy Ugandan adults: a phase 1, open-label, dose-escalation clinical trial. Lancet Infect Dis. 2023 Dec;23(12):1408-1417. doi: 10.1016/S1473-3099(23)00344-4. Epub 2023 Aug 3. PMID 37544326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the Makerere University-Walter Reed Project (MUWRP), Makerere University, in Kampala, Uganda.
Period: Overall Study
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU)
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2
Not completed — Moved from Area | 0 | 2

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 0 | 5 | 5
  21-30 years | 11 | 11 | 22
  31-40 years | 6 | 2 | 8
  41-50 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 9 | 10
  Male | 19 | 11 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  RACE: Black or African-American | 20 | 20 | 40
  ETHNICITY: Non-Hispanic/Latino | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Uganda | 20 | 20 | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.4 (3.5) | 23.7 (4.4) | 23.6 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms for 7 Days After the cAd3-EBO S Vaccine Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after the study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Incidence cAd3-EBO S Vaccine (1x10^10 PU and 1x10^11 PU): Dose groups included adults who received a single dose of cAd3-EBO S vaccine at either 1x10^10 PU or 1x10^11 PU
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) | Overall Incidence cAd3-EBO S Vaccine (1x10^10 PU and 1x10^11 PU)
Number analyzed (Participants) | 20 | 20 | 40
Participants
  Pain: None | 3 | 3 | 6
  Pain: Mild | 16 | 9 | 25
  Pain: Moderate | 1 | 8 | 9
  Pain: Severe | 0 | 0 | 0
  Swelling: None | 20 | 16 | 36
  Swelling: Mild | 0 | 3 | 3
  Swelling: Moderate | 0 | 1 | 1
  Swelling: Severe | 0 | 0 | 0
  Redness: None | 20 | 19 | 39
  Redness: Mild | 0 | 1 | 1
  Redness: Moderate | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0
  Any Local Symptom: None | 3 | 2 | 5
  Any Local Symptom: Mild | 16 | 10 | 26
  Any Local Symptom: Moderate | 1 | 8 | 9
  Any Local Symptom: Severe | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms for 7 Days After the cAd3-EBO S Vaccine Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after the study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. The majority of the reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007. The Division of AIDS AE Grading Table, Corrected Version 2.1 was used to grade reported events of joint pain (arthralgia).
Time Frame: 7 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) | Overall Incidence cAd3-EBO S Vaccine (1x10^10 PU and 1x10^11 PU)
Number analyzed (Participants) | 20 | 20 | 40
Participants
  Unusually Tired/Feeling Unwell (Malaise): None | 9 | 2 | 11
  Unusually Tired/Feeling Unwell (Malaise): Mild | 9 | 8 | 17
  Unusually Tired/Feeling Unwell (Malaise): Moderate | 2 | 10 | 12
  Unusually Tired/Feeling Unwell (Malaise): Severe | 0 | 0 | 0
  Muscle Aches (Myalgia): None | 15 | 13 | 28
  Muscle Aches (Myalgia): Mild | 5 | 5 | 10
  Muscle Aches (Myalgia): Moderate | 0 | 2 | 2
  Muscle Aches (Myalgia): Severe | 0 | 0 | 0
  Headache: None | 11 | 3 | 14
  Headache: Mild | 8 | 6 | 14
  Headache: Moderate | 1 | 11 | 12
  Headache: Severe | 0 | 0 | 0
  Chills: None | 18 | 9 | 27
  Chills: Mild | 2 | 3 | 5
  Chills: Moderate | 0 | 8 | 8
  Chills: Severe | 0 | 0 | 0
  Nausea: None | 17 | 10 | 27
  Nausea: Mild | 3 | 5 | 8
  Nausea: Moderate | 0 | 5 | 5
  Nausea: Severe | 0 | 0 | 0
  Temperature (Fever): None | 20 | 17 | 37
  Temperature (Fever): Mild | 0 | 0 | 0
  Temperature (Fever): Moderate | 0 | 2 | 2
  Temperature (Fever): Severe | 0 | 1 | 1
  Joint Pain (Arthralgia): None | 17 | 9 | 26
  Joint Pain (Arthralgia): Mild | 3 | 6 | 9
  Joint Pain (Arthralgia): Moderate | 0 | 5 | 5
  Joint Pain (Arthralgia): Severe | 0 | 0 | 0
  Any Systemic Symptom: None | 4 | 1 | 5
  Any Systemic Symptom: Mild | 13 | 3 | 16
  Any Systemic Symptom: Moderate | 3 | 15 | 18
  Any Systemic Symptom: Severe | 0 | 1 | 1

3. Primary Outcome: Total Number of Participants Reporting Any Reactogenicity Signs and Symptoms for 7 Days After the cAd3-EBO S Vaccine Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after the study product administration.
Time Frame: 7 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) | Overall Incidence cAd3-EBO S Vaccine (1x10^10 PU and 1x10^11 PU)
Number analyzed (Participants) | 20 | 20 | 40
Participants
  Total Number of Participants who had Any Local Reactogenicity Signs and Symptoms | 17 | 18 | 35
  Total Number of Participants who had Any Systemic Reactogenicity Signs and Symptoms | 16 | 19 | 35

4. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety
Description: Any abnormal laboratory results recorded as unsolicited AEs are summarized. Labs included hematology (hemoglobin, hemoglobin change from baseline, hematocrit percent, mean corpuscular volume (MCV), platelets, and white blood cell (WBC), red blood cell (RBC) and lymphocyte counts) and chemistry (alanine aminotransferase (ALT) and creatinine). Complete blood count (CBC) with total lymphocyte count results were collected at screening (≤ 56 days before enrollment), Day 0 prior to study product administration (baseline), Day 3, and Weeks 2, 4, 8 and 24. Creatinine and ALT results were collected at screening, Day 0, Day 3 and Weeks 2, 4 and 8. Institutional laboratory normal ranges as well as the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials, modified from FDA Guidance-September 2007 were used. Neutrophil results were not collected in the study database but were captured in the subject's laboratory results documentation.
Time Frame: Through 48 weeks after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) | Overall Incidence cAd3-EBO S Vaccine (1x10^10 PU and 1x10^11 PU)
Number analyzed (Participants) | 20 | 20 | 40
Participants
  ALT | 1 | 1 | 2
  WBC Count | 1 | 1 | 2
  Neutrophil Count | 1 | 2 | 3
  Hemoglobin | 0 | 0 | 0
  Hemoglobin change from baseline | 0 | 0 | 0
  Hematocrit percent | 0 | 0 | 0
  Mean corpuscular volume (MCV) | 0 | 0 | 0
  Platelets | 0 | 0 | 0
  RBC Count | 0 | 0 | 0
  Lymphocyte Count | 0 | 0 | 0
  Creatinine | 0 | 0 | 0
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 3 | 4 | 7

5. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs)
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the study product administration through the visit scheduled for 28 days after study product administration. At other time periods greater than 28 days after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module), and new chronic medical conditions that required ongoing medical management were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Through 28 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) | Overall Incidence cAd3-EBO S Vaccine (1x10^10 PU and 1x10^11 PU)
Number analyzed (Participants) | 20 | 20 | 40
Participants
  Related to Study Product | 2 | 3 | 5
  Unrelated to Study Product | 12 | 10 | 22
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 14 | 13 | 27

6. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs were recorded from receipt of the study product administration through the last expected study visit at Week 48. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Through 48 weeks after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) | Overall Incidence cAd3-EBO S Vaccine (1x10^10 PU and 1x10^11 PU)
Number analyzed (Participants) | 20 | 20 | 40
Participants
  Related to Study Product | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0
  Total Number of Participants who had an SAE | 0 | 0 | 0

7. Secondary Outcome: Geometric Mean Titers of Antibodies to the Recombinant Chimpanzee Adenovirus Serotype 3 (cAd3) Vector at 28 Days After the cAd3-EBO S Vaccine Administration
Description: Vaccine-induced, cAd3-specific antibody responses as measured by neutralization assay. Participant blood samples were tested for cAd3-specific neutralizing activity, prior to and following vaccination, using a luciferase reporter gene virus neutralization assay as previously described (Clin Vaccine Immunol 2014; 21:783-6, References Section).
Time Frame: Through 28 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: 90% neutralization titer
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU)
Number analyzed (Participants) | 20 | 20
90% neutralization titer
  Week 0 (Baseline, Pre-Administration) | 63.4 [34.6 to 116.2] | 34.3 [17.4 to 67.6]
  Week 4 (28 Days After Product Administration) | 225.2 [134.5 to 376.9] | 170.4 [77.1 to 377.0]

8. Secondary Outcome: Percentage of Participants With a Positive Ebola-Specific Antibody Response After the cAd3-EBO S Vaccine Administration
Description: A positive response is defined as a significant increase in the ELISA titer post vaccination (Week 4) compared to baseline. For each participant, a t-test was performed to compare the post vaccination titers versus those at baseline. A participant is defined as a positive responder if the one-sided t-test has a p-value < 0.05.
Time Frame: Through 28 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU)
Number analyzed (Participants) | 20 | 20
Percentage of participants | 85 [62 to 97] | 85 [62 to 97]
Statistical Analysis 1: Comparison: Group 1: cAd3-EBO S Vaccine (1x10^10 PU) vs Group 2: cAd3-EBO S Vaccine (1x10^11 PU); Statistical testing was performed within group and not between groups. Positivity for an individual was determined if there was a significant (p-value<0.05) increase (one-sided test) in the ELISA titers at week 4 when compared to those at baseline. For each participant a t-test was performed to compare the triplicate baseline titers to their triplicate week 4 titers. The proportion of positive responses and associated Clopper-Pearson 95% was calculated within group; Test type: Other — t-tests were only employed to determine which individuals were responders. Response rates with 95% Clopper-Pearson confidence intervals were reported within group; p = 0.05, t-test, 1 sided — The p-value was not adjusted for multiple comparisons and was only used to assess whether participants had a positive response or not; This test was only used to determine whether participants were positive responders or not; For each participant, a positive response was defined as a significant increase in ELISA titer post vaccination (Week 4) from baseline (Week 0). Within each participant, a t-test is performed to compare the triplicate readings (replicates 1-3) post vaccination versus the triplicate readings at baseline. A participant is defined as a positive responder if one-sided t-test has p-value < 0.05. The proportion of responders and associated 95% Clopper-Pearson Confidence Intervals were calculated

9. Secondary Outcome: Baseline-subtracted Geometric Mean Titers of cAd3-EBO S Antibodies After the cAd3-EBO S Vaccine Administration
Description: Baseline (Day 0)-subtracted geometric mean titer (GMT) was calculated along with 95% confidence intervals at Week 4 for each dose group.
Time Frame: Through 28 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU)
Number analyzed (Participants) | 20 | 20
titer | 124.9 [77.4 to 201.5] | 448.7 [249.0 to 808.7]

10. Secondary Outcome: Percentage of Participants With Positive Ebola-specific T Cell Responses After the cAd3-EBO S Vaccine Administration
Description: T cell response was measured by Intracellular Cytokine Staining (ICS) assays using Peripheral Blood Mononuclear Cells (PBMCs) at 4 weeks after vaccination. The percentage of participants with T cell responses with Clopper-Pearson 95% Confidence Intervals are presented. Positivity is defined as a response over calculated thresholds determined by the trial statistician.
Time Frame: Through 28 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU)
Number analyzed (Participants) | 20 | 20
Percentage of participants
  Percentage of Participants who produced at least one CD4 cytokine | 60 [36 to 81] | 86 [57 to 98]
  Percentage of Participants who produced at least one CD8 cytokine | 30 [12 to 54] | 29 [8 to 58]

11. Secondary Outcome: Magnitude of T Cell Response as a Percentage of EBO S-specific T Cell Subset After the cAd3-EBO S Vaccine Administration
Description: Median and interquartile ranges presented for percentage of EBO S-specific CD4 and CD8 memory T cells based on cytokine production at Week 4 for each dose group.
Time Frame: Through 28 days after study product administration
Population: All participants who received the cAd3-EBO S vaccine.
Measure: Median (Inter-Quartile Range); unit: Percentage of EBO S T cell subset
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU)
Number analyzed (Participants) | 20 | 20
Percentage of EBO S T cell subset
  CD4 T cells | 0.04 [0.02 to 0.05] | 0.08 [0.06 to 0.13]
  CD8 T cells | 0.04 [0.02 to 0.06] | 0.06 [0.03 to 0.14]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after the study product administration. Unsolicited AEs were recorded from receipt of the study product administration through the visit scheduled for 28 days after study product administration. At other time periods greater than 28 days after the study product administration, only serious AEs (SAEs), and new chronic medical conditions that required ongoing medical management were recorded through the last study visit.
Description: All AEs recorded on the study were reported. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment are reported for participants who received study product and had safety data collected following the product administration. Data represent the number and percentage of participants experiencing the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 19/20 | 19/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: cAd3-EBO S Vaccine (1x10^10 PU) (N=20) | Group 2: cAd3-EBO S Vaccine (1x10^11 PU) (N=20)
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Genital infection (Infections and infestations) | 0 | 2
Malaria (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Systemic viral infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Administration site pain (General disorders) | 17 | 17
Administration site swelling (General disorders) | 0 | 4
Administration site erythema (General disorders) | 0 | 1
Malaise (General disorders) | 11 | 18 — Unusually Tired/Feeling Unwell
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 7 — Muscle Aches
Headache (Nervous system disorders) | 9 | 17
Chills (General disorders) | 2 | 11
Nausea (Gastrointestinal disorders) | 3 | 10
Pyrexia (General disorders) | 0 | 3 — Fever
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 11 — Joint Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04041570/Prot_SAP_ICF_000.pdf